CLINICAL TRIAL: NCT06958341
Title: Registry for Patients With Antibody-mediated Neuroimmunological Diseases
Brief Title: Neuroimmunology Registry and Biobank
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Ulm (Other)
Responsible Party: Principal Investigator, Markus Schuelke, M.D., Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA2_121_17
Record Dates: First submitted 2025-04-14; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Encephalopathy; Psychosis; Impaired Consciousness; Epilepsy; Movement Disorders; Motor Neuropathy; Spasticity; Ataxia
Keywords: neuroimmunological diseases; cerebrospinal fluid; cell-based assay; tissue-based assay
MeSH Terms: conditions — Brain Diseases; Psychotic Disorders; Epilepsy; Movement Disorders; Neuritis; Muscle Spasticity; Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cerebrospinal fluid (CSF) samples stored at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with suspected neuroimmunological disease: patients with suspected neuroimmunological disease in whom a lumbar puncture is indicated for routine clinical work-up and for treatment decisions

SUMMARY:
A variety of antineuronal antibodies have been detected in the cerebrospinal fluid (CSF) of patients with neurological diseases. This raises the question of whether these antibodies are disease-specific or merely an epiphenomenon of inflammatory processes in the brain.

The registry was established with the following objectives: [1] Are antineuronal antibodies much more common than previously thought in various neurological disorders for which the etiology has not yet been elucidated? [2] Can further correlations, such as those between HSV infection and NMDA receptor autoimmunity, be identified? [3] Are these antibodies mainly non-specific epiphenomena or are they crucial for the pathogenesis? [4] What is the clinical course of patients with antineuronal antibodies and their response to therapy? These questions will be addressed in a broad immunohistological screening of a large number of CSF samples and a clinical database of patients with neurological disorders.

DETAILED DESCRIPTION:
The hypothesis that autoimmunity is a driving force behind many neurological diseases has become an established view in adult and pediatric neurology. This is particularly true for diseases of the central nervous system that are mediated by or at least associated with autoantibodies against neuronal surface antigens, the group of "autoimmune encephalitis".

This group of diseases has become increasingly important in adult neurology over the past 15 years and is now gaining importance in pediatric neurology. Since the first description of a fulminant encephalitis with autoantibodies against the N-methyl-D-aspartate (NMDA) receptor in 2007, researchers and physicians are beginning to understand that many patients worldwide with encephalopathy or epileptic and psychiatric symptoms may be suffering from previously unrecognized but treatable autoimmune diseases. As a result, the new field of "autoimmune encephalitis" has been established and new diagnostic tools are being developed. Despite a rapidly growing list of disease entities - now ranging from relatively common diagnoses such as anti-NMDA receptor, anti-α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) receptor, or anti-leucine-rich glioma-inactivated 1 (LGI1) receptor encephalitis to rare entities caused by antibodies against the metabotropic glutamate receptor 5 (mGuR5) - the field of autoimmune encephalitis is still in its infancy. The field of autoimmune encephalitis continues to evolve.

A better understanding of autoimmune encephalitis could improve the chances of treatment and even cure for many patients with previously unexplained diagnoses. This is especially true for antibody-negative autoimmune encephalitis and rare syndromes with only suspected autoantibody associations, such as corea minor and other autoimmune movement disorders, as well as ataxias, opsoclonus-myoclonus syndrome, antibody-associated motor neuronopathies, and juvenile amyotrophic lateral sclerosis (ALS). The goal of this registry is to gain new insights into the etiology of autoimmune encephalitis and non-encephalitic overlap syndromes and to investigate the role of neuronal autoantibodies in these and other neurological diseases.

The investigators will enroll patients with suspected neurologic autoimmune diseases into the database. The database will record their medical history, cardinal symptoms of the current disease, diagnostic results with emphasis on CSF analysis and imaging, as well as final diagnosis, therapy, and disease course. Residual CSF samples from lumbar punctures performed as part of the routine diagnostic workup are collected, cataloged, and stored in a CSF biobank.

The following methods are used to detect and characterize anti-neuronal antibodies: [1] highly sensitive immunofluorescence staining of fresh mouse brain (tissue-based assay, TBA), [2] immunoprecipitation from mouse brain homogenates and analysis of bound proteins by mass spectrometry, [3] flow cytometric methods (FACS, fluorescence-activated cell sorting and cell sorting), isolation and cloning of specific monoclonal autoantibodies from B-cells and plasma cells, and functional characterization studies.

ELIGIBILITY:
Inclusion Criteria:

1. Differential diagnosis: suspected neuroimmunological disease in which a lumbar puncture is indicated for further diagnosis and treatment decision
2. Individuals with unclear clinical diagnosis where additional CSF is to be collected for isolation of B cells and production of monoclonal antibodies. The clinical condition of the patients and his/her compliance have to allow an extra 2-3 ml of CSF to be collected.
3. Age: all age groups
4. Gender: patients of both sexes will be included

Exclusion criteria:

[1] Withdrawal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neurological disease in which a lumbar puncture is indicated for further diagnosis and treatment decision
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Screening for a panel of anti-neuronal antibodies via commercial assays | at recruitment
  The investigators use this commercial test battery to identify whether the CSF of the patients contains known anti-neuronal antibodies. The tests will be perfromed by Euroimmune (Lübeck, Germany). If positive, the result will be the kind of the antibody and its titer.
Screening for unknown anti-neuronal antibodies via immunofluorescence staining on fresh mouse brain (tissue-based assay, TBA) | at recruitment
  The tissue-based assay is a non-specific screening method for anti-neuronal antibodies. The investigators stain freshly cryosectioned mouse brain with patient cerebrospinal fluid at various dilutions and counterstain the sample with fluorescently labelled anti-human IgG antibodies. The sample is then imaged using fluorescence microscopy. The recorded measure will be the presence and quality of a characteristic staining pattern (cell population stained by the patient CSF) or its absence.
Determination of the molecular weight of the antibody target | at recruitment
  If the tissue based assay (TBA) is positive for a cell surface signal, the investigators will use Western blot to determine the molecular weight after staining mouse brain homogenates with patient CSF and secondary anti human anti-IgG antibodies
CSF cell count | at recruitment
  Counting and differentiating the cells found in the patient's CSF. Cell number given as "cell number per microliter". The cell type will ge given as "mononuclear cells" or "polymorph-nuclear cells"
CSF protein | at recruitment
  Measuring the protein content in the patient's CSF. The result will be given as "mg protein per ml CSF".
CSF albumin | at recruitment
  Measuring the albumin content in the patient's CSF. The result will be given as "mg albumin per ml CSF".
CSF glucose | at recruitment
  Measuring the glucose content in the patient's CSF. The result will be given as "mg glucose per liter CSF".
CSF lactate | at recruitment
  Measuring the lactate content in the patient's CSF. The result will be given as "mg lactate per liter CSF".
CSF IgG | at recruitment
  Measuring the total IgG content in the patient's CSF. The result will be given as "mg IgG per liter CSF".
CSF oligoclonal bands | at recruitment
  An electrophoresis of the patient CSF and subsequent Coomassie staining will reveal oligoclonal bande in the patient's CSF. As a result the investigators record the "presence" or "absence" of oligoclonal bands

SECONDARY OUTCOMES:
Basic clinical data | at recruitment, month 1, month 3, month 6, month 12, year 2, year 3, year 4, year 5
  The investigators will record age, height, weight, and ask about the presence of fever, weight loss, and positive findings on the internal and neurological clinical examination.
Duration from symptom onset to diagnosis | at recruitment
  The investigators will record the time delay between the occurrence of the first symptoms and the establishmen of the diagnosis. The results will be recorded as "number of days"
Assessment of the severity of ataxia | at recruitment, month 1, month 3, month 6, month 12, year 2, year 3, year 4, year 5
  The severity of the ataxia will be quantified using the Scale for the Assessment and Rating of Ataxia (SARA). The SARA score ranges between 0 (no ataxia) and 40 (most severe ataxia).
Assessment for the severity of psychiatric symptoms | at recruitment, month 1, month 3, month 6, month 12, year 2, year 3, year 4, year 5
  The severity of psychiatric symptoms, especially depression, will be quantified with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a mulitpurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Interpretation of results: minimal symptoms (5-9), minor depression (10-14), major depression (15-19), severe major depression (20-27)
Assessment of the severity of motor symptoms | at recruitment, month 1, month 3, month 6, month 12, year 2, year 3, year 4, year 5
  The Motor Function Measure (MFM) is a quantitative scale designed to describe the motor abilities of people with neuromuscular disorders. The MFM32 consists of 32 items that are scored between 0 (unable to initiate the task) and 3 (fully able to perform the task). Items fall into one of three different dimensions: Standing and transfers (D1), axial and proximal mobility (D2) and distal motor ability (D3).The raw sum score of the 32 items (maximum 96) is converted to a 0-100 scale. 100 represents full motor function.
Start and end and kind of immunotherapy | Follow-up of 5 years
  The investigators will record the date of initiation and end of the immune therapy and the kind of therapy administered.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Nikolaus, MD, Principal Investigator — Charite - Universitaetsmedizin Berlin; Tumani Hayrettin, MD, Principal Investigator — University of Ulm; Maximilian Wiesenfarth, MD, Principal Investigator — University of Ulm
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin
  - Universität Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No
The investigators do not have written consent for the sharing of individual patient data. Publication is only possible in anonymized and aggregated form.

REFERENCES:
- [Background] Kreye J, Wright SK, van Casteren A, Stoffler L, Machule ML, Reincke SM, Nikolaus M, van Hoof S, Sanchez-Sendin E, Homeyer MA, Cordero Gomez C, Kornau HC, Schmitz D, Kaindl AM, Boehm-Sturm P, Mueller S, Wilson MA, Upadhya MA, Dhangar DR, Greenhill S, Woodhall G, Turko P, Vida I, Garner CC, Wickel J, Geis C, Fukata Y, Fukata M, Pruss H. Encephalitis patient-derived monoclonal GABAA receptor antibodies cause epileptic seizures. J Exp Med. 2021 Nov 1;218(11):e20210012. doi: 10.1084/jem.20210012. Epub 2021 Sep 21. PMID 34546336
- [Background] Nikolaus M, Kuhne F, Tietze A, Thumfart J, Kempf C, Gratopp A, Knierim E, Bittigau P, Kaindl AM. Modified Zipper Method, a Promising Treatment Option in Severe Pediatric Immune-Mediated Neurologic Disorders. J Child Neurol. 2022 May;37(6):505-516. doi: 10.1177/08830738221089476. Epub 2022 Apr 18. PMID 35435761
- [Background] Nikolaus M, Koch A, Stenzel W, Elezkurtaj S, Sahm F, Tietze A, Stoffler L, Kreye J, Hernaiz Driever P, Thomale UW, Kaindl AM, Schuelke M, Knierim E. Atypical NMDA receptor expression in a diffuse astrocytoma, MYB- or MYBL1-altered as a trigger for autoimmune encephalitis. Acta Neuropathol. 2022 Aug;144(2):385-389. doi: 10.1007/s00401-022-02447-y. Epub 2022 Jun 21. No abstract available. PMID 35727368
- [Background] Schnell S, Knierim E, Bittigau P, Kreye J, Hauptmann K, Hundsdoerfer P, Morales-Gonzalez S, Schuelke M, Nikolaus M. Hodgkin Lymphoma Cell Lines and Tissues Express mGluR5: A Potential Link to Ophelia Syndrome and Paraneoplastic Neurological Disease. Cells. 2023 Feb 13;12(4):606. doi: 10.3390/cells12040606. PMID 36831273
- [Background] Wilpert NM, de Almeida Marcelino AL, Knierim E, Incoronato P, Sanchez-Sendin E, Staudacher O, Drenckhahn A, Bittigau P, Kreye J, Pruss H, Schuelke M, Kuhn AA, Kaindl AM, Nikolaus M. Pediatric de novo movement disorders and ataxia in the context of SARS-CoV-2. J Neurol. 2023 Oct;270(10):4593-4607. doi: 10.1007/s00415-023-11853-5. Epub 2023 Jul 29. PMID 37515734
- [Background] Viezens I, Knierim E, Deubzer HE, Hauptmann K, Fassbender J, Morales-Gonzalez S, Kaindl AM, Schuelke M, Nikolaus M. Expression of mGluR5 in Pediatric Hodgkin and Non-Hodgkin lymphoma-A Comparative Analysis of Immunohistochemical and Clinical Findings Regarding the Association between Tumor and Paraneoplastic Neurological Disease. Cancers (Basel). 2024 Jul 4;16(13):2452. doi: 10.3390/cancers16132452. PMID 39001514
- [Background] Wendel EM, Tibussek D, Barisic N, Bertolini A, Panzer A, Chang P, Geis T, Knierim E, Nikolaus M, Nosadini M, Sartori S, Schoene-Bake JC, Yilmaz D, Reindl M, Pakeerathan T, Ayzenberg I, Rostasy K. Children with MOG-IgG positive bilateral optic neuritis misdiagnosed as fulminant idiopathic intracranial hypertension. Mult Scler Relat Disord. 2025 Jan;93:106205. doi: 10.1016/j.msard.2024.106205. Epub 2024 Dec 15. PMID 39675122
- [Background] Cramer P, Nikolaus M, Loos S, Denecke J, Knierim E, Muller D, Weber LT, Taylan C, Thumfart J. Immunoadsorption is equally effective as plasma exchange in paediatric neuroimmunological disorders - A retrospective multicentre study. Eur J Paediatr Neurol. 2025 Jan;54:58-63. doi: 10.1016/j.ejpn.2024.12.005. Epub 2024 Dec 21. PMID 39752845
- [Background] Kauth F, Bertolini A, Wendel EM, Koukou G, Naggar IE, Chung J, Baumann M, Schodl C, Lechner C, Bigi S, Blaschek A, Hengstler JG, Schimmel M, Nosadini M, Sartori S, Puthenparampil M, Van's Gravesande KS, Drenckhahn A, Nikolaus M, Kauffmann B, Thiels C, Hausler MG, Eckenweiler M, Karenfort M, Marina AD, Selek A, Oncel I, Kornek B, Reindl M, Rostasy K. Characterization of children with early onset pediatric multiple sclerosis. Eur J Paediatr Neurol. 2025 Jan;54:113-120. doi: 10.1016/j.ejpn.2025.01.006. Epub 2025 Jan 23. PMID 39879856